CLINICAL TRIAL: NCT01661790
Title: Open-labeled, Randomized, Multicenter Phase III Study of Adjuvant Chemotherapy Comparing Bevacizumab Plus Cisplatin With Cisplatin Regimen in Malignant Pleural Effusion of Advanced Stage Non-Small-Cell Lung Cancer Patients
Brief Title: Intrapleural Bevacizumab and Cisplatin Therapy for Malignant Pleural Effusion Caused by Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, DuNan, director of oncology department in PLA 304 hospital, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLA304DN-001
Record Dates: First submitted 2012-07-25; First posted 2012-08-10 (Estimated); Results first posted 2015-03-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Malignant Pleural Effusion
Keywords: Bevacizumab;; non-small cell lung cancer;; malignant pleural effusion;; intrapleural administration
MeSH Terms: conditions — Pleural Effusion, Malignant; Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab & Cisplatin (Experimental): Bevacizumab 300mg plus Cisplatin 30mg by intrapleural given every two weeks
  Interventions: Drug: Bevacizumab; Drug: Cisplatin
- Cisplatin (Active Comparator): Cisplatin 30mg by intrapleural given every two weeks
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab300mg&Cispltin30mg by intrapleural administration of each 2 week
  Other Names: Avastin
  Arms: Bevacizumab & Cisplatin
Drug: Cisplatin — Cisplatin 30mg,intrapleural administration,each 2 week

SUMMARY:
To determine the efficacy and Safety of intrapleural Bevacizumab and cisplatin as a treatment for malignant pleural effusions (MPE) in patients with non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced recurrent or progressive NSCLC proven cytohistologically
* Karnofsky performance status (KPS) ≥60
* Life expectancy ≥ 2 months
* No history of severe diseases of major organs including liver, heart, and kidney
* No previous intrapleural therapy
* Written informed consent

Exclusion Criteria:

* Active thoracic cavity or systemic bleeding
* Active pleural or systemic infection.
* Known sensitivity to Bevacizumab or Cisplatin
* Refusal to participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-08; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nan Du, Principal Investigator — PLA 304 hospital
Locations (1):
- PLA 304 hospital, Beijing, Beijing Municipality, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab & Cisplatin: Bevacizumab 300mg plus Cisplatin 30mg by intrapleural given every two weeks
  Bevacizumab: Bevacizumab300mg&Cisplatin 30mg by intrapleural administration of each 2 week
  Cisplatin: Cisplatin 30mg,intrapleural administration,each 2 week
- Cisplatin: Cisplatin 30mg by intrapleural given every two weeks
  Cisplatin: Cisplatin 30mg,intrapleural administration,Q2W
Period: Overall Study
Arm/Group | Bevacizumab & Cisplatin | Cisplatin
Started | 36 | 36
Completed | 36 | 34
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Bevacizumab & Cisplatin: Bevacizumab 300mg plus Cisplatin 30mg by intrapleural given every two weeks
  Bevacizumab: Bevacizumab300mg&Cisplatin 30mg by intrapleural administration of each 2 week
  Cisplatin: Cisplatin 30mg,intrapleural administration,Q2W
- Total: Total of all reporting groups
Arm/Group | Bevacizumab & Cisplatin | Cisplatin | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 20 | 18 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With "Complete Response" and "Partial Response"
Description: Response assessed by type-B ultrasonic tests; Complete remission (CR) was considered when the accumulated fluid had disappeared and was stable for at least four weeks; partial remission (PR) was considered when >50% of the accumulated fluid had disappeared, symptoms had improved, and the remaining fluid had failed to increase for at least four weeks; The total efficiency ORR was calculated by taking the sum of CR+PR
Time Frame: from randomization, This treatment was given every two weeks,responses were made by biweekly
Measure: Number; unit: participants
Arm/Group | Bevacizumab & Cisplatin | Cisplatin
Number analyzed (Participants) | 36 | 34
participants
  CR | 17 | 2
  PR | 13 | 15

2. Secondary Outcome: Median Progression Free Survival (PFS)
Time Frame: baseline to biweekly,until disease progression
Reporting Status: Not Posted

3. Secondary Outcome: Overall Survival (OS)
Time Frame: randomization to four weeks,until death
Reporting Status: Not Posted

4. Secondary Outcome: Adverse Reactions
Time Frame: Up to 1 month after the last treatment
Reporting Status: Not Posted

5. Secondary Outcome: Qualify of Life (QoL)
Time Frame: baseline to biweekly,until death
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Quantitative RT-PCR(Reverse Transcription-Polymerase Chain Reaction) for VEGF-A(Vascular Endothelial Growth Factor A)
Time Frame: before intrapleural administration
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Bevacizumab & Cisplatin | Cisplatin
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 24/36 | 22/36
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab & Cisplatin (N=36) | Cisplatin (N=36)
Leucocytopenia (Blood and lymphatic system disorders) | 24 (24) | 22 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes